CLINICAL TRIAL: NCT07190105
Title: Impact of Vagal Approaches on Symptomatology in Long COVID Participants
Brief Title: Vagal Approaches on Long COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leidos Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LDOS-25-001; MCDC2015-003 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-09-22; First posted 2025-09-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Long COVID Symptoms
Keywords: COVID; Long COVID; Covid-19; Fitbit; Sonic Augmentation Technology (SAT); Electrical Vagus Nerve Stimulator; General Wellness Product; Autonomic Nervous System; Vagus Nerve; Sonocea; Truvaga
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sonocea Sonic Augmentation Technology (SAT) General Wellness Product (Experimental): Participants enrolled in this arm will listen to a sound-based approach, delivered via headphones through a smartphone application. The session participants will listen to consists of structured music soundscapes that have been standardized in format, intensity, and duration for research purposes.
  Interventions: Other: Sonocea Sonic Augmentation Technology (SAT)
- Truvaga Electrical Vagus Nerve Stimulator General Wellness Product (Experimental): Participants enrolled in this arm will use the Truvaga Electrical Vagus Nerve Stimulator general wellness product, which sends gentle electrical signals through the skin to stimulate the vagus nerve on the neck.
  Interventions: Other: Truvaga Electrical Vagus Nerve Stimulator
- Sonocea SAT + Truvaga Electrical Vagus Nerve Stimulator General Wellness Products (Experimental): Participants enrolled in this arm will use both the Sonocea SAT and Truvaga Electrical Vagus Nerve Stimulator general wellness products.
  Interventions: Other: Sonocea Sonic Augmentation Technology (SAT); Other: Truvaga Electrical Vagus Nerve Stimulator
- Control (No Intervention) (No Intervention): Participants enrolled in this arm will not use either wellness product.

INTERVENTIONS:
Other: Sonocea Sonic Augmentation Technology (SAT) — The Sonocea Sonic Augmentation Technology (SAT) is a sound-based approach delivered via headphones through a smartphone application. The approach uses music soundscapes that have been standardized in format, intensity and duration.
  Arms: Sonocea SAT + Truvaga Electrical Vagus Nerve Stimulator General Wellness Products; Sonocea Sonic Augmentation Technology (SAT) General Wellness Product
Other: Truvaga Electrical Vagus Nerve Stimulator — The Truvaga Electrical Vagus Nerve Stimulator is a general wellness product that sends gentle electrical signals through the skin to stimulate the vagus nerve on the neck.
  Arms: Sonocea SAT + Truvaga Electrical Vagus Nerve Stimulator General Wellness Products; Truvaga Electrical Vagus Nerve Stimulator General Wellness Product

SUMMARY:
The purpose of this study is to explore whether two general wellness products, alone or combined, can support individuals experiencing Long COVID symptoms. Both wellness products stimulate the vagus nerve - a nerve that helps regulate stress, relaxation, mood, breathing, heart rate, inflammation, and digestion.

The investigators will use a Fitbit to track participants' health measurements including, but not limited to, activity, heart rate, and heart rate variability, and participants will be asked to complete surveys about their experience. This information will be collected into a repository where participants can share their experiences with Long COVID symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Tested positive by any test for acute COVID-19 and/or have ICD-10 code for COVID-19 in their electronic health records (EHR)
2. Any patient having the ICD-10 code for post-acute sequelae of COVID-19 (PASC) within their EHR, or any patient who has evidence of a Long COVID clinic visit within their EHR
3. Have persistent COVID-19 symptoms 3 months following resolution of acute COVID-19 infection as indicated by a negative COVID-19 test
4. Self-identified as having Long COVID based on symptomology:

   a. Symptoms must include any combination of the following: (ICD-10 codes shown):
   * Shortness of breath (R06.02, R06.00, or R06.09)
   * Fatigue (R53.83, or R53.82)
   * Cognitive impairment (G31.84 or R41.9)
   * Mental, Behavioral, and Neurodevelopmental disorders (F01-F99)
   * Postural orthostatic tachycardia syndrome (POTS) (I49.8)
5. Participants must have auditory headphones; over the ear headphones or earbuds
6. Participants must be at least 18 years of age, inclusive, at the time of signing the informed consent
7. Capable of understanding and providing signed informed consent
8. Participants must have a smart phone
9. Reliable access to internet via browser installed on a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2025-10-27 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-8 (PHQ-8) | Week 0, Week 4 and Week 8
  The PHQ-8 is a gold-standard screening tool for major depressive disorder, endorsed by the CDC and WHO, with strong criterion validity and sensitivity to clinical change.
Generalized Anxiety Disorder-7 (GAD-7) | Week 0, Week 4 and Week 8
  The GAD-7 captures both somatic and cognitive components of generalized anxiety. Extensively used in both clinical and epidemiological contexts, the GAD-7 shows excellent internal consistency (α > 0.90) and convergent validity with clinician-administered diagnostic tools.
PTSD Checklist for DSM-5 Short Form (Abbreviated PCL-5) | Week 0, Week 4 and Week 8
  The Abbreviated PCL-5 captures re-experiencing, avoidance, hyperarousal, and mood alterations. The Abbreviated PCL-5 is validated across diverse populations and is widely used in both military and civilian trauma research. It is recommended by the National Center for PTSD.
Symptom Burden Questionnaire - Long COVID (SBQ-LC) | Week 0, Week 4 and Week 8
  The SBQ-LC measures the intensity and impact of Long COVID symptoms, offering key insight into the ongoing symptom burden experienced. The SBQ-LC demonstrates strong psychometric properties with high internal consistency across subscales and good convergent validity with established measures of symptom severity and functional impairment. It has been validated across diverse Long COVID populations in multiple clinical settings.
Body Perception Questionnaire (BPQ) | Week 0, Week 4 and Week 8
  The BPQ assesses self-reported autonomic reactivity and has been used in a range of international neural, behavioral, and clinical studies and translated into several languages. It has been corroborated with sensor-based measures of autonomic function.
Benefits Scale | Weekly
  The Benefits Scale assesses biobehavioral state, including the ability to quiet thoughts, awareness of bodily rhythms, breathing, muscular relaxation, physical pain levels, and emotional states such as peacefulness, relaxation, anxiety, irritability, feeling overwhelmed, worry about the future, and vulnerability.
Sleep Metrics | Weekly
  The investigators will use the sleep categories of accumulated minutes of deep sleep, REM sleep, light sleep, and wakefulness during the night to provide us with sleep architecture.
Resting Heart Rate | Weekly
  Monitoring resting heart rate will allow us to assess whether SAT and Truvaga Electrical Vagus Nerve Stimulator are effective in lowering the elevated resting heart rate often observed in Long COVID patients via parasympathetic stimulation.
Steps | Weekly
  Monitoring steps will allow us to assess whether SAT and Truvaga Electrical Vagus Nerve Stimulator are associated with an increase in average daily steps, which may indicate enhanced functional capacity or reduced fatigue.
Breathing Rate | Weekly
  This measurement captures a user's average breaths per minute during sleep.
Heart Rate Variability (HRV) | Weekly
  Heart rate variability (HRV) is a widely recognized biomarker for autonomic nervous system regulation. Long COVID is commonly associated with reduced HRV, reflecting autonomic nervous system dysregulation. Lower HRV in these patients has been linked to greater symptom burden.
Cardio Score (VO2 Max) | Weekly
  Tracking changes in estimated aerobic capacity can help evaluate whether approaches are improving cardiovascular function and exercise tolerance over time.
SpO2 | Weekly
  SpO2 measures blood oxygen saturation levels, indicating how well oxygen is being transported throughout the body.
Active Zone Minutes | Weekly
  Active Zone Minutes are a measure of time spent in elevated heart rate zones, including Fat Burn, Cardio, and Peak zones.

OTHER OUTCOMES:
The Adverse and Traumatic Experiences Scale (ATES) | Week 0
  ATES captures developmental and lifetime adversity that may impact vagal tone and neuroception. The ATES will allow us to examine the effectiveness of SAT and the Electrical Vagus Nerve Stimulator in individuals who report being impacted by their adversity histories.
Brain Body Center Sensory Scale (BBCSS) | Week 0, Week 4 and Week 8
  The BBCSS assesses sensory processing difficulties that may reflect underlying autonomic dysfunction.
Purpose in Life (PIL-SF) | Week 0, Week 4 and Week 8
  The PIL-SF measures existential meaning, motivational vitality, and psychological presence.
Neuroception of Psychological Safety Scale (NPSS) | Week 0, Week 4 and Week 8
  The NPSS evaluates subjective experiences of social safety/co-regulation and physiological regulation.
Sonic Augmentation Technology (SAT) Support Needs Scale | Week 0
  This tool enables tailored interpretation of individual differences in responsivity to Sonic Augmentation Technology and vagus nerve stimulation, particularly in populations with heightened neurophysiological sensitivity or neurodivergent traits.

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual, Frederick, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Results from the study will be analyzed and reported in accordance with the protocol and applicable regulations. Additionally, findings may be shared in presentations, publications, or other formats as determined by the study team and stakeholders.